CLINICAL TRIAL: NCT00281684
Title: A Multi-centre, Randomised, Single Blind, Placebo Controlled, Parallel Group Study to Examine the Effect of Single Doses of SB-705498, a TRPV1 Receptor Antagonist, on Pain Following Third Molar Tooth Extraction
Brief Title: SB-705498 Dental Pain Study After Tooth Extraction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: VRA105345
Record Dates: First submitted 2006-01-23; First posted 2006-01-25 (Estimated); Results first posted 2019-01-28 (Actual); Last update posted 2019-01-28 (Actual); Status verified 2017-09

CONDITIONS: Toothache
Keywords: Acute Pain; Dental Pain; Vanilloid; VR1; TRPV1; Inflammation
MeSH Terms: conditions — Toothache; Acute Pain; Inflammation | interventions — SB 705498; acetaminophen, codeine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Experimental): Eligible participants received a single dose of SB705498 matching placebo capsules (4 placebo capsules) via oral route and were followed up to a maximum of 14 days.
  Interventions: Drug: Placebo
- SB705498 400 mg (Experimental): Eligible participants received a single dose of SB705498 400 milligram (mg) capsules (2 x 200 mg capsules plus 2 placebo capsules) via oral route and were followed up to a maximum of 14 days.
  Interventions: Drug: SB705498 400 mg
- SB705498 1000 mg (Experimental): Eligible participants received a single dose of SB705498 1000 mg capsules (2 x 200 mg capsules plus 2 x 300 mg capsules) via oral route and were followed up to a maximum of 14 days.
  Interventions: Drug: SB705498 1000 mg
- Co-Codamol (Experimental): Eligible participants received a single dose of Co-codamol capsules (2 x Paracetamol Ph Eur 500 mg, codeine phosphate hemihydrate Ph Eur 12.8 mg plus two placebo capsules) via oral route and were followed up to a maximum of 14 days.
  Interventions: Drug: Co-Codamol

INTERVENTIONS:
Drug: SB705498 400 mg — SB705498 400 mg
  Arms: SB705498 400 mg
Drug: SB705498 1000 mg — SB705498 1000 mg
  Arms: SB705498 1000 mg
Drug: Placebo — Placebo
  Arms: Placebo
Drug: Co-Codamol — Co-Codamol
  Arms: Co-Codamol

SUMMARY:
This clinical trial is a multi centre, randomised, single-blind, parallel group, placebo-controlled, single oral dose study with a positive control arm. Patients previously scheduled for 3rd molar tooth extraction, who are otherwise healthy, will be recruited. Upon completion of surgery, e.g. prior to established pain, patients will be randomised to treatment (SB-706598, placebo or co-codamol) and dosed with the study medication

ELIGIBILITY:
Inclusion criteria:

* Female or male subjects aged 18 to 50. Women may be of child bearing potential or of non-child bearing potential. Women of child bearing potential must use an effective method of contraception (see below).
* Females of non-child bearing potential are defined as:
* Post-menopausal females, being amenorrhoeic for at least 2 years with an appropriate clinical profile, e.g., age appropriate, history of vasomotor symptoms. However, if indicated this should be confirmed by oestradiol and FSH levels consistent with menopause (according to local laboratory ranges).
* Pre-menopausal females with a documented hysterectomy (medical report verification) and/or bilateral oophorectomy. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
* Subject is healthy. Healthy subjects are defined as individuals who are not taking any regular medication and are free from clinically significant illness or disease as determined by their medical history (including family history), physical examination, 12-lead ECG, Holter monitor, laboratory studies, and other tests specified in this protocol.
* Subject is scheduled for outpatient surgical removal of up to four third molar teeth under local anesthesia. At least one third molar tooth must be a fully or partially impacted in the mandible requiring bone removal;
* Subject agrees not to take analgesics other than protocol defined rescue analgesics during treatment (up to 24 hrs post dose)
* Subject has the ability to read, comprehend, and record information required by protocol;
* Subject is willing and able to provide signed and dated written informed consent prior to study participation.

Exclusion criteria:

* Subject has a history or presence of significant organ disease or mental illness;
* Subject has been exposed to analgesics other than aspirin (including prescription and over the counter NSAIDs or COX-2 inhibitors) within 24 hours prior to the start of surgery;
* Subject is unable to refrain from alcohol, psychoactive drugs, and sedatives including sleeping preparations (e.g . benzodiazepines) within 24 hours prior to the start of surgery and for the duration of their participation in the study
* Following screening (and 24 h Holter ECG) the subject has a significant abnormality that, in the opinion of the investigator makes them unsuitable for the study.
* Subject with a known allergy to or judged by the investigator not to be a suitable candidate for ibuprofen or co-codamol therapy based on medical history, concomitant medications, and concurrent systemic disease as described in the product labeling, e.g., peptic ulcer disease, angioedema, bronchospastic reactivity (e.g., asthma), rhinitis and nasal polyps induced by aspirin or other NSAIDs;
* The subject had a history of drug or alcohol abuse, or had a positive pre-study urine drug / alcohol breath screen. Abuse of alcohol is defined as an average weekly intake of greater than 21 units or an average daily intake of greater than three units for males and intake greater than 14 units per week or an average daily intake of greater than two units for females. One unit is equivalent to a half-pint (220 mL) of beer or one (25 mL) measure of spirits or one glass (125 mL) of wine.
* Subject has participated, or is participating in, a clinical study in which they have been exposed to an investigational drug or device during the past 30 days;
* Subject has donated blood (450 mL or more) within the previous month.
* Male subjects only:
* An unwillingness of male subjects to abstain from sexual intercourse with pregnant or lactating women from the time of the first dose of study medication until five half-lives following administration of the last dose of study medication.
* An unwillingness of the male subject to use a condom/spermicide in addition to having their female partner use another form of contraception such as IUD, diaphragm with spermicide, oral contraceptives, injectable progesterone, subdermal implants or a tubal ligation if the woman could become pregnant from the time of the first dose of study medication until 84 days following administration of the last dose of study medication.
* Female subjects of child bearing potential:
* Female subjects who are pregnant, breast feeding, or have a positive serum pregnancy test or a positive urine pregnancy test either at screening or pre-dose on each dosing session.
* An unwillingness of the female subject to use an appropriate form of contraception. Appropriate forms of contraception are defined as:
* Abstinence - The lifestyle of the female should be such that there is complete abstinence from intercourse from at least the commencement of their last normal period prior to the first dose of study medication and to continue until the first normal period (defined as normal for the woman, both in terms of duration and quantity of menses) after treatment or 15 days after the last dose of medication, whichever is the longest.
* One of the following methods is acceptable as the sole method of contraception if there is indisputable data that it is >99% effective otherwise it should be used with a barrier method (condom or occlusive cap {diaphragm or cervical/vault caps} used with spermicidal foam/gel/film/cream/suppository):
* Established use of oral, injected or implanted hormonal methods of contraception from at least the commencement of their last normal period prior to the first dose of study medication. Subjects using hormonal contraception should use a barrier method in addition from the first dose of study medication until their next normal period following the end of the study.
* Documented tubal ligation.
* Documented placement of an intrauterine device (IUD) or intrauterine system (IUS).
* Male partner sterilisation (vasectomy) prior to the female subject's entry into the study and is the sole partner for that female subject.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 145 (Actual)
Dates: Start 2005-12-07 (Actual); Primary Completion 2007-10-03 (Actual); Study Completion 2007-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- GSK Investigational Site, Verona, Veneto, Italy
- GSK Investigational Site, Seoul, South Korea
- United Kingdom (3):
  - GSK Investigational Site, Croydon, Surrey
  - GSK Investigational Site, Leeds
  - GSK Investigational Site, Manchester

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 3 centers in the United Kingdom, 1 center in Korea, Republic of and 1 center in Italy from 07 December 2005 to 03 October 2007. A total of 145 participants were enrolled into the study.
Pre-assignment Details: Participants already scheduled for 3rd molar tooth extraction, who were otherwise healthy, were recruited for this study. As soon as reasonably possible after completion of tooth extraction (but within 1 hour), participants were randomized to treatment and dosed with the study medication whilst local anesthetic was still active.
Groups:
- Co-Codamol: Eligible participants received a single dose of Co-codamol capsules (2 x Paracetamol European Pharmacopoeia [Ph Eur] 500 mg, codeine phosphate hemihydrate Ph Eur 12.8 mg plus two placebo capsules) via oral route and were followed up to a maximum of 14 days.
Period: Overall Study
Arm/Group | Placebo | SB705498 400 mg | SB705498 1000 mg | Co-Codamol
Started | 37 | 36 | 34 | 38
Completed | 36 | 36 | 33 | 38
Not Completed | 1 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- SB705498 400 mg: Eligible participants received a single dose of SB705498 400 mg capsules (2 x 200 mg capsules plus 2 placebo capsules) via oral route and were followed up to a maximum of 14 days.
- Total: Total of all reporting groups
Arm/Group | Placebo | SB705498 400 mg | SB705498 1000 mg | Co-Codamol | Total
Number analyzed (Participants) | 37 | 36 | 34 | 38 | 145
Age, Continuous [Mean (Standard Deviation); unit: Years] | 27.5 (7.37) | 27.0 (6.45) | 26.0 (7.26) | 27.0 (6.36) | 26.9 (6.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 18 | 20 | 19 | 76
  Male | 18 | 18 | 14 | 19 | 69
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 11 | 5 | 15 | 12 | 43
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 1
  Black or African American | 1 | 1 | 1 | 2 | 5
  White | 25 | 29 | 18 | 23 | 95
  More than one race | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean of Pain Intensity Based on the Visual Analogue Scale (VAS)
Description: Pain intensity was assessed using VAS. These assessments were then summarized to give a weighted mean score. The VAS was a subjective assessment of post-operative pain intensity. The participants rated the pain intensity at the time of assessment by marking a line on a 100 millimeter (mm) (0 to 100 mm) long scale. A line placed on the extreme left (0 mm) indicated no pain and extreme right (100 mm) indicated worst pain imaginable. This scale has no subscales. Only those participants available at the specified time points were analyzed.
Time Frame: Up to 10 hours post-dose
Population: The Intent-to-Treat (ITT) population which comprised of all participants randomized to treatment, who took the study medication and who had at least one post-dose assessment. The ITT population did not include participants who took rescue medication or withdrew within the first 120 minutes after administration of study medication.
Measure: Least Squares Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Placebo | SB705498 400 mg | SB705498 1000 mg | Co-Codamol
Number analyzed (Participants) | 35 | 34 | 32 | 36
Scores on a Scale | 37.45 (22.474) | 34.95 (26.076) | 38.84 (22.869) | 17.15 (26.094)

2. Secondary Outcome: Change From Baseline in the Pain Intensity Based on the Verbal Rating Scale (VRS) up to 10 Hours Post Baseline
Description: Pain intensity was assessed using VRS. Participants also used a 4-point categorical VRS for the subjective assessment of postoperative pain. The score and it corresponding intensity was such that 0= no pain, 1= mild, 2= moderate and 3= severe. The VRS was collected as an independent measure of the participant's pain and was not prospectively correlated to the study participant's numerical score (number of millimeters) on the VAS. Participants were provided with a worksheet with a list of adjectives to read and they were asked to select the word by checking the box that best described their level of pain. The number associated with the adjective chosen by the participant constituted the pain intensity. Baseline (Day 1) value was the value obtained immediately prior to administration of study drug. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values.
Time Frame: Up to 10 hours post Baseline (Day 1)
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Placebo | SB705498 400 mg | SB705498 1000 mg | Co-Codamol
Number analyzed (Participants) | 37 | 34 | 33 | 38
Scores on a Scale
  Pre-dose: number analyzed (Participants) | 35 | 34 | 32 | 36
  Pre-dose | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  1 hour post-randomization: number analyzed (Participants) | 35 | 34 | 32 | 36
  1 hour post-randomization | 0.3 (0.51) | 0.3 (0.80) | 0.6 (0.62) | 0.3 (0.51)
  2 hour post-randomization: number analyzed (Participants) | 35 | 34 | 32 | 36
  2 hour post-randomization | 1.3 (0.89) | 1.1 (1.05) | 1.3 (0.90) | 0.9 (0.87)
  3 hour post-randomization: number analyzed (Participants) | 23 | 18 | 17 | 29
  3 hour post-randomization | 1.3 (0.75) | 1.0 (0.91) | 1.4 (0.79) | 1.0 (1.07)
  4 hour post-randomization: number analyzed (Participants) | 18 | 15 | 13 | 25
  4 hour post-randomization | 1.3 (0.77) | 1.1 (1.03) | 1.2 (0.90) | 1.0 (1.06)
  5 hour post-randomization: number analyzed (Participants) | 16 | 11 | 11 | 22
  5 hour post-randomization | 1.2 (0.83) | 0.9 (0.83) | 0.8 (0.60) | 1.1 (0.99)
  6 hour post-randomization: number analyzed (Participants) | 13 | 11 | 9 | 17
  6 hour post-randomization | 1.1 (0.76) | 1.0 (0.89) | 0.9 (0.60) | 1.0 (1.06)
  7 hour post-randomization: number analyzed (Participants) | 12 | 11 | 8 | 15
  7 hour post-randomization | 1.2 (0.83) | 1.1 (0.83) | 0.9 (0.64) | 0.8 (1.08)
  8 hour post-randomization: number analyzed (Participants) | 12 | 10 | 8 | 13
  8 hour post-randomization | 1.0 (0.74) | 0.9 (0.88) | 0.8 (0.71) | 0.8 (1.28)
  9 hour post-randomization: number analyzed (Participants) | 11 | 8 | 8 | 12
  9 hour post-randomization | 1.0 (0.77) | 0.6 (0.74) | 0.8 (0.71) | 0.7 (1.23)
  10 hour post-randomization: number analyzed (Participants) | 11 | 8 | 7 | 10
  10 hour post-randomization | 1.1 (0.83) | 0.8 (1.04) | 0.6 (0.53) | 0.5 (1.18)

3. Secondary Outcome: Change From Baseline in the Pain Intensity Based on the VAS up to 10 Hours Post-Baseline
Description: Pain intensity was assessed using VAS. The VAS was a subjective assessment of post-operative pain intensity. The participants rated the pain intensity at the time of the assessment by marking a line on a 100 millimeter (mm) (0 to 100 mm) long scale. A line placed on the extreme left (0 mm) indicated no pain and extreme right (100 mm) indicated worst pain imaginable. This scale has no subscales. The Baseline (Day 1) value was the value obtained immediately prior to administration of study drug. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values.
Time Frame: Baseline (Day 1) to 10 hours post Baseline
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Placebo | SB705498 400 mg | SB705498 1000 mg | Co-Codamol
Number analyzed (Participants) | 37 | 34 | 33 | 38
Scores on a Scale
  1 hour post randomization: number analyzed (Participants) | 35 | 34 | 32 | 36
  1 hour post randomization | 4.7 (9.12) | 8.0 (17.66) | 10.0 (16.55) | 4.6 (9.40)
  2 hour post randomization: number analyzed (Participants) | 35 | 34 | 32 | 36
  2 hour post randomization | 27.8 (22.02) | 26.9 (30.74) | 34.6 (24.72) | 15.2 (25.76)
  3 hour post randomization: number analyzed (Participants) | 23 | 18 | 17 | 29
  3 hour post randomization | 27.1 (17.10) | 13.7 (18.96) | 39.0 (25.52) | 15.7 (26.09)
  4 hour post randomization: number analyzed (Participants) | 18 | 15 | 13 | 25
  4 hour post randomization | 29.6 (20.16) | 18.6 (23.22) | 36.4 (26.07) | 16.8 (25.08)
  5 hour post randomization: number analyzed (Participants) | 16 | 11 | 11 | 22
  5 hour post randomization | 25.8 (18.98) | 11.5 (23.56) | 25.8 (20.96) | 14.3 (21.50)
  6 hour post randomization: number analyzed (Participants) | 13 | 11 | 9 | 17
  6 hour post randomization | 25.9 (19.00) | 13.8 (24.91) | 28.3 (21.19) | 10.5 (26.51)
  7 hour post randomization: number analyzed (Participants) | 12 | 11 | 8 | 15
  7 hour post randomization | 25.9 (21.55) | 15.7 (24.64) | 25.6 (19.65) | 8.0 (28.17)
  8 hour post randomization: number analyzed (Participants) | 12 | 10 | 8 | 13
  8 hour post randomization | 19.5 (18.59) | 12.2 (25.28) | 24.0 (18.88) | 6.5 (28.92)
  9 hour post randomization: number analyzed (Participants) | 11 | 8 | 8 | 12
  9 hour post randomization | 17.0 (16.94) | 6.6 (19.81) | 19.6 (15.03) | 10.3 (32.63)
  10 hour post randomization: number analyzed (Participants) | 11 | 8 | 7 | 10
  10 hour post randomization | 17.1 (20.52) | 7.3 (20.27) | 17.0 (15.47) | 7.2 (25.19)

4. Secondary Outcome: Elapsed Time From Study Drug Administration to Rescue Analgesic Request
Description: Duration of Analgesic Effect (Time to First Rescue medication from study drug administration) is presented. Ibuprofen 400 mg was provided as rescue medication to be taken as required. The time when the rescue medication was administered was recorded on the case report form.
Time Frame: Within 24 hours of administration of study drug
Population: ITT Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | Placebo | SB705498 400 mg | SB705498 1000 mg | Co-Codamol
Number analyzed (Participants) | 37 | 34 | 33 | 38
Hours | 5.13 [2.08 to 10.33] | 4.27 [2.02 to 19.70] | 3.12 [2.12 to 11.08] | 6.88 [2.28 to 11.92]

5. Secondary Outcome: Number of Participants With Different Global Evaluation or Overall Impression of Study Medication Use and at 10 and 24 Hours Post Randomization
Description: Participants subjectively assessed their overall impression (global evaluation) of the study medication using a 4-point categorical scale, where 1= poor, 2= fair, 3= good and 4= excellent. Participants were provided with a list of adjectives and were asked to select the word by checking the box that best rated the study medication that they received for pain relief. The number associated with the adjective chosen by the participant constituted the global evaluation score. The study coordinator or designee transcribed the number corresponding to the selected adjective onto the case report form. The Global Evaluation was completed prior to receiving the first rescue medication, at 10 hours post-dose and prior to discharge from the unit.
Time Frame: Prior to first rescue medication use and at 10 and 24 hours post randomization
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SB705498 400 mg | SB705498 1000 mg | Co-Codamol
Number analyzed (Participants) | 37 | 34 | 33 | 38
Participants
  Pre-rescue: Poor | 9 | 7 | 10 | 8
  Pre-rescue: Fair | 9 | 10 | 6 | 9
  Pre-rescue: Good | 8 | 6 | 6 | 12
  Pre-rescue: Excellent | 0 | 1 | 0 | 2
  At 10 hour post-randomization: Poor | 0 | 0 | 0 | 0
  At 10 hour post-randomization: Fair | 0 | 0 | 0 | 0
  At 10 hour post-randomization: Good | 0 | 0 | 1 | 0
  At 10 hour post-randomization: Excellent | 0 | 0 | 0 | 0
  At 24 hour post-randomization: Poor | 11 | 9 | 14 | 9
  At 24 hour post-randomization: Fair | 10 | 9 | 6 | 11
  At 24 hour post-randomization: Good | 9 | 12 | 9 | 13
  At 24 hour post-randomization: Excellent | 3 | 4 | 3 | 3

6. Secondary Outcome: VAS Mean Pain Scores From the Time of Rescue Medication up to 10 Hours Post Randomization
Description: Pain intensity was assessed using VAS. VAS was a subjective assessment of post-operative pain intensity. Participants rated the pain intensity at the time of assessment by marking a line on a 100 mm (0 to 100 mm) long scale. A line placed on extreme left, i.e., 0 mm indicated no pain and extreme right that is 100 mm indicated worst pain imaginable. This scale has no subscales.
Time Frame: From the time of rescue medication to 10 hours post randomization
Population: ITT Population. Only those participants who used rescue medication were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Placebo | SB705498 400 mg | SB705498 1000 mg | Co-Codamol
Number analyzed (Participants) | 37 | 34 | 33 | 38
Scores on a Scale
  3 hour post-randomization: number analyzed (Participants) | 12 | 16 | 16 | 7
  3 hour post-randomization | 74.7 (18.68) | 70.1 (17.87) | 61.7 (26.50) | 70.9 (22.57)
  4 hour post-randomization: number analyzed (Participants) | 17 | 19 | 20 | 11
  4 hour post-randomization | 69.4 (19.14) | 64.9 (22.12) | 59.2 (26.64) | 65.5 (26.05)
  5 hour post-randomization: number analyzed (Participants) | 19 | 23 | 22 | 14
  5 hour post-randomization | 66.4 (20.25) | 61.9 (21.83) | 59.8 (26.53) | 63.5 (27.58)
  6 hour post-randomization: number analyzed (Participants) | 21 | 23 | 24 | 19
  6 hour post-randomization | 63.9 (20.79) | 61.9 (21.83) | 59.3 (25.65) | 56.2 (27.23)
  7 hour post-randomization: number analyzed (Participants) | 22 | 23 | 25 | 21
  7 hour post-randomization | 64.9 (20.83) | 61.9 (21.83) | 60.4 (25.67) | 55.1 (26.03)
  8 hour post-randomization: number analyzed (Participants) | 22 | 24 | 25 | 24
  8 hour post-randomization | 64.9 (20.83) | 61.5 (21.43) | 60.4 (25.67) | 55.8 (24.56)
  9 hour post-randomization: number analyzed (Participants) | 23 | 26 | 24 | 25
  9 hour post-randomization | 65.7 (20.70) | 59.9 (21.31) | 60.6 (26.20) | 55.0 (24.40)
  10 hour post-randomization: number analyzed (Participants) | 23 | 26 | 26 | 27
  10 hour post-randomization | 65.7 (20.70) | 59.9 (21.31) | 59.9 (25.29) | 53.7 (24.29)

7. Secondary Outcome: Number of Participants Requiring Rescue Medication Over Time
Description: Ibuprofen 400 mg was provided as rescue medication to be taken as required. The time that rescue medication was administered was recorded on the case report form. Number of participants requiring rescue medication up to 10 hour post-dose are presented.
Time Frame: Up to 10 hour post-dose
Population: ITT Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SB705498 400 mg | SB705498 1000 mg | Co-Codamol
Number analyzed (Participants) | 37 | 34 | 33 | 38
Participants
  1 hour post-dose | 0 | 0 | 0 | 0
  2 hour post-dose | 0 | 0 | 0 | 0
  3 hour post-dose | 12 | 16 | 16 | 7
  4 hour post-dose | 17 | 19 | 20 | 11
  5 hour post-dose | 19 | 23 | 22 | 14
  6 hour post-dose | 21 | 23 | 24 | 19
  7 hour post-dose | 22 | 23 | 25 | 21
  8 hour post-dose | 22 | 24 | 25 | 24
  9 hour post-dose | 23 | 26 | 24 | 25
  10 hour post-dose | 23 | 26 | 26 | 27

8. Secondary Outcome: Number of Participants From First Rescue Medication Use to Second Rescue Analgesic Request
Description: Ibuprofen 400 mg was provided as rescue medication to be taken as required. The time that rescue medication was administered was recorded on the case report form. Number of participants using the second rescue medication from the time the first rescue medication was used are presented.
Time Frame: From first dose of rescue medication to second dose of rescue medication
Population: ITT Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SB705498 400 mg | SB705498 1000 mg | Co-Codamol
Number analyzed (Participants) | 37 | 34 | 33 | 38
Participants | 6 | 5 | 10 | 9

9. Secondary Outcome: Number of Participants With Adverse Events (AE) Over Time
Description: AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. For marketed medicinal products, this also includes failure to produce expected benefits (i.e., lack of efficacy), abuse or misuse.
Time Frame: Up to Follow-up (28 days)
Population: The Safety population which comprised of all participants who were randomized and took at least one capsule of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SB705498 400 mg | SB705498 1000 mg | Co-Codamol
Number analyzed (Participants) | 37 | 36 | 34 | 38
Participants | 16 | 10 | 14 | 14

10. Secondary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Findings
Description: ECGs were recorded with the participant lying supine, having rested in this position for at least 5 minutes before each recording. Full 12 lead ECGs were recorded using an ECG device that automatically calculated the heart rate and measured PR, QRS, RR, QT and QT, QT corrected by Bazett's formula (QTcB) and QT corrected by Fridericia's formula (QTcF) intervals. Paper ECG traces were recorded at a standard paper speed of 25 millimeter/second and gain of 1mVolt/10 millimeter, using 2.5x4 format with lead II rhythm strip. Cardiac intervals were checked by a physician and then transcribed into the case report form. Number of participants with abnormal (not clinically significant [NCS] and clinically significant [CS]) ECG findings are presented.
Time Frame: 28 days
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SB705498 400 mg | SB705498 1000 mg | Co-Codamol
Number analyzed (Participants) | 37 | 36 | 34 | 38
Participants
  Pre-dose, Abnormal-NCS | 9 | 7 | 14 | 10
  Pre-dose, Abnormal-CS | 0 | 0 | 0 | 0
  2 hour post-dose, Abnormal-NCS | 16 | 10 | 15 | 7
  2 hour post-dose, Abnormal-CS | 0 | 0 | 0 | 0
  4 hour post-dose, Abnormal-NCS | 8 | 9 | 15 | 7
  4 hour post-dose, Abnormal-CS | 0 | 0 | 0 | 0
  6 hour post-dose, Abnormal-NCS | 4 | 9 | 8 | 9
  6 hour post-dose, Abnormal-CS | 0 | 0 | 0 | 0
  8 hour post-dose, Abnormal-NCS | 7 | 9 | 11 | 6
  8 hour post-dose, Abnormal-CS | 0 | 0 | 0 | 0
  10 hour post-dose, Abnormal-NCS | 8 | 11 | 13 | 8
  10 hour post-dose, Abnormal-CS | 0 | 0 | 0 | 0
  24 hour post-dose, Abnormal-NCS | 7 | 12 | 10 | 8
  24 hour post-dose, Abnormal-CS | 0 | 0 | 0 | 0

11. Secondary Outcome: Number of Participants With Second Degree Atrioventricular Block Over 24 Hours by Holter Tape
Description: Continuous ambulatory Holter ECG monitoring was performed for a 24-hour period at screening (Day -14 to Day -1) and from pre-dose (post surgery) to approximately 20 hours post-randomization. Number of participants with second degree atrioventricular block over 24 hours by Holter tape are presented.
Time Frame: Up to 24 hours post-dose
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SB705498 400 mg | SB705498 1000 mg | Co-Codamol
Number analyzed (Participants) | 37 | 36 | 34 | 38
Participants | 0 | 0 | 1 | 1

12. Secondary Outcome: Change From Baseline for Vital Signs- Diastolic Blood Pressure (DBP) and Systolic Blood Pressure (SBP)
Description: Supine SBP and DBP measurements were performed with the participant in a supine position after the participant has rested for at least 5 minutes. Assessment was completed pre-dose and then at 2, 4, 6, 8, 10 and discharge (approximately 24 hour) post randomization. Baseline (Day 1) value was the value obtained immediately prior to administration of study drug. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values.
Time Frame: Baseline (Day 1) to 24 hours post Baseline
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Placebo | SB705498 400 mg | SB705498 1000 mg | Co-Codamol
Number analyzed (Participants) | 37 | 36 | 34 | 38
Millimeters of mercury (mmHg)
  DBP: 2 hour post-randomization | 7.62 (8.388) | 5.94 (9.411) | 5.62 (7.758) | 2.84 (8.952)
  DBP: 4 hour post-randomization: number analyzed (Participants) | 37 | 36 | 33 | 38
  DBP: 4 hour post-randomization | 3.11 (7.770) | 2.36 (7.772) | 4.06 (8.489) | 2.16 (8.106)
  DBP: 6 hour post-randomization: number analyzed (Participants) | 36 | 36 | 34 | 38
  DBP: 6 hour post-randomization | 4.03 (7.129) | -0.33 (8.384) | -2.18 (6.930) | 2.50 (7.783)
  DBP: 8 hour post-randomization: number analyzed (Participants) | 36 | 36 | 34 | 38
  DBP: 8 hour post-randomization | 1.44 (6.631) | 1.25 (8.005) | -1.50 (7.712) | -0.08 (7.691)
  DBP: 10 hour post-randomization: number analyzed (Participants) | 36 | 36 | 34 | 38
  DBP: 10 hour post-randomization | 0.67 (6.612) | -0.25 (6.971) | -0.91 (6.824) | -0.87 (8.217)
  DBP: 24 hour post-randomization: number analyzed (Participants) | 36 | 36 | 34 | 38
  DBP: 24 hour post-randomization | -0.61 (6.677) | -1.97 (7.113) | -1.74 (6.426) | -2.32 (7.956)
  SBP: 2 hour post-randomization | 8.08 (10.087) | 5.25 (9.488) | 7.18 (10.641) | 2.39 (10.640)
  SBP: 4 hour post-randomization: number analyzed (Participants) | 37 | 36 | 33 | 38
  SBP: 4 hour post-randomization | 5.08 (10.133) | 3.97 (9.782) | 7.09 (11.145) | 4.42 (11.377)
  SBP: 6 hour post-randomization: number analyzed (Participants) | 36 | 36 | 34 | 38
  SBP: 6 hour post-randomization | 5.06 (10.656) | 0.11 (10.717) | 1.21 (9.380) | 2.84 (9.474)
  SBP: 8 hour post-randomization: number analyzed (Participants) | 36 | 36 | 34 | 38
  SBP: 8 hour post-randomization | 2.08 (9.533) | 1.28 (10.859) | -0.65 (7.908) | 0.08 (8.556)
  SBP: 10 hour post-randomization: number analyzed (Participants) | 36 | 36 | 34 | 38
  SBP: 10 hour post-randomization | 2.31 (11.887) | -0.44 (8.433) | 1.06 (9.335) | 2.18 (8.693)
  SBP: 24 hour post-randomization: number analyzed (Participants) | 36 | 36 | 34 | 38
  SBP: 24 hour post-randomization | 0.58 (8.897) | -1.03 (9.238) | -0.32 (8.138) | -0.13 (8.777)

13. Secondary Outcome: Change From Baseline for Vital Signs-Body Temperature
Description: Tympanic temperature was assessed at screening, pre-dose and then at 2, 4, 6, 8, 10 and discharge (approximately 24 hours) post-Baseline. Temperature was also recorded at the follow-up visit. The Baseline (Day 1) value was the value obtained immediately prior to administration of study drug. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values.
Time Frame: Baseline (Day 1) to 24 hours post Baseline
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | Placebo | SB705498 400 mg | SB705498 1000 mg | Co-Codamol
Number analyzed (Participants) | 37 | 36 | 34 | 38
Degree Celsius
  2 hour post randomization: number analyzed (Participants) | 21 | 14 | 34 | 23
  2 hour post randomization | 0.17 (0.345) | 0.28 (0.635) | 0.47 (0.399) | 0.07 (0.446)
  4 hour post randomization: number analyzed (Participants) | 21 | 14 | 33 | 23
  4 hour post randomization | 0.27 (0.402) | 0.49 (0.604) | 0.74 (0.446) | 0.24 (0.404)
  6 hour post randomization: number analyzed (Participants) | 20 | 14 | 34 | 23
  6 hour post randomization | 0.47 (0.423) | 0.59 (0.708) | 0.75 (0.481) | 0.41 (0.487)
  8 hour post randomization: number analyzed (Participants) | 21 | 14 | 34 | 23
  8 hour post randomization | 0.50 (0.525) | 0.33 (0.699) | 0.67 (0.546) | 0.45 (0.654)
  10 hour post randomization: number analyzed (Participants) | 21 | 14 | 34 | 23
  10 hour post randomization | 0.43 (0.569) | 0.28 (0.598) | 0.46 (0.532) | 0.32 (0.625)
  24 hour post randomization: number analyzed (Participants) | 20 | 14 | 34 | 23
  24 hour post randomization | 0.26 (0.421) | 0.37 (0.809) | 0.45 (0.618) | 0.34 (0.624)

14. Secondary Outcome: Number of Participants With Clinical Chemistry/ Hematology Values/ Serum Hormones Values of Potential Clinical Concern
Description: Hematology parameters included hemoglobin, packed cell volume, mean cell hemoglobin, mean cell hemoglobin concentration, red blood cell count, white blood cell (WBC) count, platelets and differential WBC count. Clinical chemistry parameters included sodium, potassium, urea, creatinine, total protein, albumin, total bilirubin, aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase, gamma glutamyl transferase (GGT), lactate dehydrogenase, calcium, magnesium, phosphate, cholesterol, high density lipoprotein cholesterol, triglycerides, glucose and creatinine kinase. Only those parameters for which at least one value of potential clinical concern was reported are presented.
Time Frame: Up to 28 days
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SB705498 400 mg | SB705498 1000 mg | Co-Codamol
Number analyzed (Participants) | 37 | 36 | 34 | 38
Participants
  Alkaline Phosphatase, High at Follow-up | 0 | 0 | 0 | 1
  Alanine Amino Transferase, High at screening | 0 | 1 | 0 | 0
  Alanine Amino Transferase, High at Follow-up | 0 | 1 | 1 | 0
  Total Bilirubin, High at screening | 2 | 1 | 0 | 6
  Total Bilirubin, High at 24 hour post-dose | 5 | 3 | 6 | 8
  Total Bilirubin, High at Follow-up | 1 | 0 | 0 | 0
  Calcium, Low at Follow-up | 1 | 0 | 0 | 0
  Creatine Kinase, High at screening | 2 | 1 | 2 | 5
  Creatine Kinase, High at 24 hour post-dose | 0 | 0 | 1 | 1
  Creatine Kinase, High at Follow-up | 0 | 1 | 1 | 2
  GGT, High at screening | 0 | 0 | 0 | 1
  GGT, High at 24 hour post-dose | 0 | 0 | 0 | 2
  GGT, High at Follow-up | 0 | 0 | 0 | 2
  Glucose, High at 24 hour post-dose | 1 | 0 | 0 | 0
  Glucose, High at Follow-up | 0 | 1 | 0 | 0
  Glucose, Low at Follow-up | 1 | 0 | 0 | 0
  Hemoglobin, Low at Follow-up | 1 | 0 | 0 | 0
  Potassium, High at screening | 0 | 1 | 0 | 0
  Potassium, High at 24 hour post-dose | 0 | 1 | 0 | 0
  Sodium, Low at Follow-up | 1 | 0 | 0 | 0
  WBC count, High at 24 hour post-dose | 0 | 0 | 0 | 2

15. Secondary Outcome: Number of Participants With Abnormal Urine Parameters
Description: Urinalysis parameters included protein, glucose, ketones, bilirubin, blood, urobilinogen, urine leukocyte esterase (ULE) test for detecting WBC (via dipstick method). The dipstick test gives results in a semi-quantitative manner, and results for urinalysis parameter of urine can be read as negative, Trace, +, ++, +++ and ++++ indicating proportional concentrations in the urine sample. The results above ++ that is ++, +++ and ++++ were reported as abnormal and the corresponding parameters were considered as abnormal parameters. Number of participants with abnormal urinalysis parameters were reported.
Time Frame: Up to 28 days
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SB705498 400 mg | SB705498 1000 mg | Co-Codamol
Number analyzed (Participants) | 37 | 36 | 34 | 38
Participants
  Urine Bilirubin, ++ | 0 | 1 | 0 | 0
  Urine Ketones, ++ | 2 | 1 | 1 | 1
  Urine Leukocyte Esterase, ++ | 2 | 7 | 3 | 3
  Urine microscop-Cellular Casts, ++ | 1 | 1 | 0 | 0
  Urine microscop-Culture, ++ | 2 | 1 | 0 | 0
  Urine Occult Blood, ++ | 1 | 2 | 2 | 2
  Urine Ketones, +++ | 0 | 3 | 1 | 1
  Urine Leukocyte Esterase, +++ | 0 | 1 | 1 | 0
  Urine microscopy-Culture, +++ | 1 | 2 | 0 | 0
  Urine Occult Blood, +++ | 4 | 3 | 3 | 2

16. Secondary Outcome: Area Under Curve (AUC)(0-rescue) and AUC(0-t) of SB705498
Description: Cannulation of the forearm vein was performed prior to surgery for serial pharmacokinetic blood sampling. The cannula was kept patent by means of a 0.9% saline lock. Blood was sampled via the intravenous cannula with 1 mL of blood being withdrawn prior to each sample and discarded. Venipuncture was allowed if necessary (e.g., cannulation failure).
Time Frame: At pre-dose on Baseline (Day 1) and at between 20-40 minutes and at 1, 1.5, 2, 3, 4, 6, 8, 10 hours post dose and at final follow-up (Day 28)
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram*hour per milliliter (ug*h/mL)
Arm/Group | SB705498 400 mg | SB705498 1000 mg
Number analyzed (Participants) | 34 | 33
Microgram*hour per milliliter (ug*h/mL)
  AUC(0-rescue): number analyzed (Participants) | 32 | 33
  AUC(0-rescue) | 1.6684 (82.462) | 2.2589 (82.989)
  AUC(0-t): number analyzed (Participants) | 32 | 33
  AUC(0-t) | 3.1467 (51.813) | 4.8338 (38.963)

17. Secondary Outcome: Plasma Concentrations: Average Concentration (C-avg) [0-rescue] and Maximum Concentration (C-max) of SB705498
Description: as for outcome 16
Time Frame: as for outcome 16
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter (ug/mL)
Arm/Group | SB705498 400 mg | SB705498 1000 mg
Number analyzed (Participants) | 32 | 33
Microgram per milliliter (ug/mL)
  C-avg (0-rescue) | 0.3387 (42.682) | 0.5472 (36.126)
  C-max | 0.5855 (43.101) | 0.8903 (41.759)

18. Secondary Outcome: Time Prior to the First Measurable Concentration (T-lag) and Time to Maximum Observed Plasma Concentration (T-max)
Description: as for outcome 16
Time Frame: At pre-dose (Baseline) and at between 20-40minutes and at 1, 1.5, 2, 3, 4, 6, 8, 10 hours post randomization and at final follow-up (Day 28)
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Median (Full Range); unit: Hour
Arm/Group | SB705498 400 mg | SB705498 1000 mg
Number analyzed (Participants) | 32 | 33
Hour
  T-lag | 0.00 [0.0 to 0.5] | 0.00 [0.0 to 0.0]
  T-max | 1.500 [1.00 to 8.15] | 1.500 [1.00 to 10.15]

ADVERSE EVENTS:
Time Frame: Up to 28 days
Description: Safety population was used for this analysis.
Arm/Group | Placebo | SB705498 400 mg | SB705498 1000 mg | Co-Codamol
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/36 | 0/34 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/36 | 0/34 | 0/38
Other Adverse Events (participants affected / at risk) | 16/37 | 10/36 | 14/34 | 14/38
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=37) | SB705498 400 mg (N=36) | SB705498 1000 mg (N=34) | Co-Codamol (N=38)
Headache (Nervous system disorders) | 5 | 1 | 5 | 4
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 3
Dizziness postural (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope vasovagal (Nervous system disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Feeling hot (General disorders) | 2 | 0 | 2 | 0
Pyrexia (General disorders) | 0 | 1 | 2 | 0
Catheter site pain (General disorders) | 1 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 1 | 0
Feeling abnormal (General disorders) | 0 | 0 | 0 | 1
Feeling cold (General disorders) | 0 | 0 | 1 | 0
Feeling of body temperature change (General disorders) | 0 | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 1 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 1 | 1
Asthenopia (Eye disorders) | 1 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 1 | 0 | 0
ACTH stimulation test (Investigations) | 0 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.